## Development and Implementation of Electronic Decision Aids for Genetic Testing in Inherited Cancer Syndromes

NCT04704193

July 18th, 2024

The analysis will be descriptive in nature. We will tabulate the responses for all survey items from all participants who completed the survey. The primary outcomes are the 6 items related to participant satisfaction with how educational information is presented in the decision aid, with each rated as poor, fair, good or excellent. The results will be summarized with count and percentage for each response category. The secondary outcome is the amount of time spent on the decision aid, which will be summarized using mean with standard deviation or median with interquartiles if the distribution is skewed.